CLINICAL TRIAL: NCT01526005
Title: Brain Nicotine Receptor Density & Response to Nicotine Patch
Status: Completed | Type: Observational
Sponsor: Brentwood Biomedical Research Institute (Other)
Responsible Party: Principal Investigator, Arthur Brody, Principal Investigator, Brentwood Biomedical Research Institute
Other Study IDs: 0015
Record Dates: First submitted 2011-08-29; First posted 2012-02-03 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active agent (nicotine patch)
  Interventions: Drug: Transdermal Nicotine Patch
- Placebo patch
  Interventions: Drug: Transdermal Placebo Patch

INTERVENTIONS:
Drug: Transdermal Nicotine Patch — 1 patch per day; dosages of 21 mg/day for 4 weeks, 14 mg/day for 2 weeks, and 7 mg/day for 2 weeks; 8 weeks total
  Groups: Active agent (nicotine patch)
Drug: Transdermal Placebo Patch — 1 patch per day; 8 weeks total
  Groups: Placebo patch

SUMMARY:
Even though the health risks and societal costs of cigarette smoking are well-known, roughly 19.8% of American adults continue to smoke. While most smokers endorse a desire to quit, very few (< 5%) will actually quit in a given year without treatment, and only about 20-25% achieve abstinence after 6 months or more of effective treatment. Therefore, there continues to be a vital need to improve outcomes for cigarette smokers seeking treatment. Current first-line medications for Tobacco Dependence include nicotine replacement therapies (such as the patch, gum, lozenge, nasal spray, and inhaler), varenicline HCl (Chantix), and bupropion HCl (Zyban), with the current standard of care in most treatment settings being to choose specific medications based primarily on availability, ease of use, and patient preference. The goal of the proposed research is to improve the delivery of smoking cessation treatment by determining if pre-treatment nicotine receptor density in cigarette smokers is associated with smoking cessation outcome with the standard nicotine patch taper. The study's main hypothesis is that cigarette smokers with less pre-treatment upregulation of nicotine receptors will have a greater likelihood of quitting smoking from a standard course of nicotine patch treatment than smokers with more up-regulation of these receptors. Positron emission tomography (PET) will be used to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult who is a tobacco dependent smoker (smokes 10-30 cigarettes per day) meeting criteria for Nicotine Dependence as defined by DSM-IV criteria
* Has the desire to quit smoking
* Ability to read, write, and give voluntary informed consent
* An exhaled CO greater than or equal to 8 ppm during the study screening visit to verify smoking status

Exclusion Criteria:

* Any history of an Axis I psychiatric diagnosis other than Nicotine Dependence (including other substance abuse/dependence and mood, anxiety, and psychotic disorders)
* Any current medication or any history of a medical condition that might affect the central nervous system at the time of scanning (e.g., current treatment with a psychotropic medication, or history of severe head trauma or epilepsy).
* Unstable cardiovascular disease, liver disease, or renal insufficiency. Routine history and physical examination will be performed at the initial screening visit to insure that participants meet study criteria
* Pregnancy (urine pregnancy tests will be obtained on all women of child-bearing potential) due to the theoretical risk of radiation exposure to the fetus. Pre-menopausal women will only be scanned during the early follicular phase (by participant report) of the menstrual cycle because hormonal levels have been shown to affect nicotine metabolism.
* Caffeine dependence, as evidenced by withdrawal symptoms temporally associated with caffeine ingestion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Tobacco dependent cigarette smokers will be recruited through newspaper and internet advertisements from populations living in the counties surrounding the West Los Angeles Veterans Affairs Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
PET scanning | 2/12-2/14
  Brain imaging used to predict response to smoking cessation treatment

CONTACTS AND LOCATIONS:
Locations (1):
- West Los Angeles Veterans Affairs Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Brody AL, Mukhin AG, Mamoun MS, Luu T, Neary M, Liang L, Shieh J, Sugar CA, Rose JE, Mandelkern MA. Brain nicotinic acetylcholine receptor availability and response to smoking cessation treatment: a randomized trial. JAMA Psychiatry. 2014 Jul 1;71(7):797-805. doi: 10.1001/jamapsychiatry.2014.138. PMID 24850280